CLINICAL TRIAL: NCT06645236
Title: Interventional IVD Study Testing DNA From Tumor Tissue Biopsies From mCRC Patients to Determine KRAS G12C Mutation Status for the Inclusion in the Amgen Clinical Trial, 20210081 for the Clinical Performance of Therascreen® KRAS RGQ PCR Kit
Brief Title: DHF-20-1839-2: Clinical Performance Study Protocol for Therascreen® KRAS RGQ PCR Kit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DHF-20-1839-2
Record Dates: First submitted 2023-12-20; First posted 2024-10-16 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Colorectal Cancer (mCRC)
Keywords: Metastatic Colorectal Cancer; therascreen; KRAS G12C; sotorasib; Clinical Performance Study; Companion Diagnostic
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clinical Performance Study Protocol for therascreen® KRAS RGQ PCR Kit (Other): The therascreen® KRAS RGQ PCR Kit functions as part of this system, using the QIAamp DSP DNA FFPE Kit as a clinical sample concentrator, the Rotor-Gene Q MDx (RGQ) instrument as the platform on which PCR is performed, and KRAS specific software for PCR analysis and result reporting. The kit contains a Positive Control (PC) and a No Template Control (NTC) which are used to determine the validity of the test.
  The therascreen® KRAS RGQ PCR Kit is a real-time qualitative PCR assay used on the Rotor-Gene Q MDx (US) instrument for the detection of seven somatic mutations in the human KRAS oncogene, using DNA extracted from formalin-fixed, paraffin-embedded (FFPE), colorectal cancer (CRC) tissue
  Interventions: Device: therascreen® KRAS RGQ PCR Kit

INTERVENTIONS:
Device: therascreen® KRAS RGQ PCR Kit — The investigational device, therascreen® KRAS RGQ PCR Kit, will be used to determine the KRAS G12C mutation status of patients during the screening period of Amgen's clinical trial (20210081)

SUMMARY:
To utilize the therascreen KRAS RGQ PCR Kit, as a screening test in Amgen's Phase 3 Clinical Study Protocol 20210081, in order to identify patients with mCRC KRAS G12C mutation positive tumors to be enrolled in the drug clinical trial. Results of the Phase 3 Amgen Study 20210081 will serve as the basis for establishing the clinical performance of the therascreen® KRAS RGQ PCR Kit as a companion diagnostic (CDx) for the identification of patients with metastatic colorectal cancer, who may benefit from treatment with sotorasib.

DETAILED DESCRIPTION:
The proposed device clinical performance study and the medicinal clinical trial will be conducted simultaneously as a combined trial according to MDCG 2022-10. The clinical trial 20210081 is a Randomized, Open-label, Active-controlled Study of Sotorasib, Panitumumab and FOLFIRI Versus FOLFIRI With or Without Bevacizumab-awwb for Treatment-naïve Subjects with Metastatic Colorectal Cancer with KRAS p.G12C Mutation (CodeBreaK 301). It is estimated that approximately 450 patients from 31 countries will be enroled based on the presence of tumor KRAS G12C mutation, detected using therascreen KRAS RGQ PCR Kit, along with other clinical trial inclusion criteria, into the Phase III clinical trial. Results from the Phase 3 Amgen Study 20210081 will be used to evaluate the clinical performance of therascreen® KRAS RGQ PCR Kit as a CDx device for identification of patients with mCRC who may benefit from treatment with sotorasib in treatment-naïve patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who consent to participate in the eligibility screen for Protocol 20210081 will have their tumor tissue tested for the presence of KRAS G12C mutation under the proposed performance study.

Exclusion Criteria:

* There is no separate inclusion and exclusion criteria for the performance study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-12-22 (Actual); Primary Completion 2030-10-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
Detection of KRAS G12C mutation status | 6 years; due to end 2030
  Detection of the KRAS G12C mutation status in DNA extracted from Formalin-Fixed Paraffin-Embedded (FFPE), CRC tissue using the therascreen KRAS RGQ PCR Kit to enrol approximately 450 KRAS G12C positive patients for clinical study protocol 20210081.
Progression Free Survival (PFS) | 6 years; due to end 2030
  The primary efficacy endpoint is progression free survival (PFS), defined as time from randomization until disease progression or death from any cause, whichever occur first as per the sotorasib clinical trial (Protocol 2021008).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, Dr., Study Director — Qiagen Manchester Limited
Locations (1):
- QIAGEN Gaithersburg, Inc, Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No